CLINICAL TRIAL: NCT00191789
Title: Neoadjuvant Administration of Gemcitabine Plus Doxorubicin Followed by Gemcitabine Plus Cisplatin in Large or Locally Advanced Operable Breast Cancer: A Phase II Study
Brief Title: Neoadjuvant Sequential Administration of Two Gemcitabine Combinations in Operable Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7117; B9E-MC-S329 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2010-07-22 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Doxorubicin; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine+Doxorubicin+Cisplatin+Surgery (Experimental): Gemcitabine: 1200 mg/m^2, intravenous (IV) day 1 and day 8 every 21 days x 4 cycles (1-4) then 1000 mg/m^2, IV, day 1 and day 8 every 21 days x 4 cycles (5-8).
  Doxorubicin: 60 mg/m^2, IV, every 21 days x 4 cycles (1-4). Cisplatin: 70 mg/m^2, IV, every 21 days x 4 cycles (5-8). Surgery follows 8 cycles of chemotherapy. Extent and type of surgery is guided by tumor size, physician and/or patient decision.
  Interventions: Drug: gemcitabine; Drug: doxorubicin; Drug: cisplatin; Procedure: surgery

INTERVENTIONS:
Drug: gemcitabine — 1200 mg/m^2, intravenous (IV) day 1 and day 8 every 21 days x 4 cycles (1-4) then 1000 mg/m^2, IV, day 1 and day 8 every 21 days x 4 cycles (5-8)
  Other Names: LY188011; Gemzar
Drug: doxorubicin — 60 mg/m^2, IV, every 21 days x 4 cycles (1-4)
Drug: cisplatin — 70 mg/m^2, IV, every 21 days x 4 cycles (5-8)
Procedure: surgery — Surgery follows 8 cycles of chemotherapy. Extent and type of surgery is guided by tumor size, physician and/or patient decision.

SUMMARY:
Gemcitabine and anthracycline combination has shown encouraging activity as neoadjuvant chemotherapy in locally advanced breast cancer. An addition of sequential gemcitabine and cisplatin, also a highly active combination in this indication, may result in improvement in pathological response and overall survival. Patients with operable breast cancer will be treated in neoadjuvant setting with gemcitabine plus doxorubicin, followed by gemcitabine plus cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast carcinoma
* No previous chemotherapy, with bidimensionally measurable locally advanced disease
* Adequate performance status (Karnofsky Performance Status [KPS] greater than or equal to 70), bone marrow reserves, hepatic, cardiac and renal functions.

Exclusion Criteria:

* Inflammatory breast cancer
* Pregnancy and Breast-feeding
* Serious concomitant disorder or infection
* Previous cancer within the last 5 years or a second primary malignancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2003-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern Time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- India (3):
  - For additional information regarding investigative sites for this clinical trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT -5 hours, EST), or speak with your personal physician., Pune, Maharashtra
  - For additional information regarding investigative sites for this clinical trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT -5 hours, EST), or speak with your personal physician., Vellore, Tamil Nadu
  - For additional information regarding investigative sites for this clinical trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT -5 hours, EST), or speak with your personal physician., Delhi

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Started | 65
Completed | 40
Not Completed | 25
Not completed — Adverse Event | 5
Not completed — Patient: Satisfactory Response | 5
Not completed — Patient/Physician: Satisfactory Response | 4
Not completed — Withdrawal by Subject | 4
Not completed — Death - Possibly Study Drug Related | 4
Not completed — Progressive Disease/Lack of Efficacy | 2
Not completed — Death - Not Study-Drug Related | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Number analyzed (Participants) | 65
Age Continuous [Median (Full Range); unit: years] | 46 [31 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Indian | 65
Region of Enrollment [Number; unit: participants]
  India | 65
Diagnosis [Number; unit: participants]
  Histopathological | 12
  Cytological | 53
Disease Stage [Number; unit: participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body).
  Stage IIA-cancer cells found in lymph nodes, or tumor is larger than 2 cm, but less than 5 cm and not in lymph nodes; Stage IIB - tumor larger than 2 cm, but less than 5 cm and in lymph nodes, or tumor larger than 5 cm but not in lymph nodes; Stage IIIA - cancer has spread to nearby tissues; Stage IIIB - cancer has spread to chestwall and/or skin, and lymph nodes near breastbone.
  participants
    Stage IIA | 3
    Stage IIB | 30
    Stage IIIA | 18
    Stage IIIB | 14
Hormone Receptor Status [Number; unit: participants] — Status of the estrogen receptors (ER) and progesterone receptors (PR). A score of Estrogen Receptor positive (ER+) means that estrogen is causing the tumor to grow and Progesterone Receptor positive (PR+) means that progesterone is causing the tumor to grow.
  participants
    ER+ / PR+ | 27
    ER+ / PR- | 8
    ER- / PR+ | 3
    ER- / PR- | 25
    No Assessment | 2
Human Epidermal Growth Factor Receptor 2 (HER-2) Status [Number; unit: participants] — Status determines if there is too much HER-2 receptor protein on the surface of the breast cancer cell. Results range from 0 (negative), 1+ (negative), 2+ (borderline) to 3+ (positive).
  participants
    0 | 27
    1+ | 8
    2+ | 2
    3+ | 19
    Not Detected | 7
    Insufficient Sample | 2
Karnofsky Performance Status Scale [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0-100 (in increments of 10), the lower the score, the worse the survival for most serious illnesses.
  participants
    100 - Normal no complaints; no evidence of disease | 9
    90 - Normal activity; minor signs of disease | 56
Menopausal Status [Number; unit: participants]
  Premenopausal | 29
  Postmenopausal | 36
Body Surface Area [Median (Full Range); unit: meters squared (m^2)] — The calculation is from the formula of DuBois and DuBois: BSA = (Weight^0.425 x Height^0.725) x 0.007184, where weight is in kilograms and height is in centimeters.
  meters squared (m^2) | 1.44 [1.19 to 1.77]
Height [Median (Full Range); unit: centimeters (cm)] | 153 [141 to 170]
Largest Lesion Size [Median (Full Range); unit: millimeters (mm)] | 30 [7.8 to 85.8]
Weight [Median (Full Range); unit: kilograms (kg)] | 57 [34 to 87]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pathological Complete Response (Pathological Complete Response Rate)
Description: Complete pathological response: No invasive tumor cells identified from sections from site of previous cancer. Require evidence corroborating prior presence of invasive cancer, which requires detection of abnormal fibroelastic breast stroma devoid of normal lobular units and contains foamy macrophages with moderate numbers of fibroblasts and mononuclear inflammatory cells. Presence of nondescript collagenised lobules or breast fibrous tissue is not evidence that tumor site has been adequately sampled and macroscopic assessment and sampling is needed until original neoplastic stroma identified.
Time Frame: tumor assessment at baseline and during surgery after eight 21-day treatment cycles
Population: Intent to treat population.
Measure: Number; unit: participants
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Number analyzed (Participants) | 65
participants | 13

2. Secondary Outcome: Summary of Deaths During Study
Time Frame: baseline through last cycle on study drug (eight 21-day cycles)
Population: Intent to treat population.
Measure: Number; unit: participants
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Number analyzed (Participants) | 65
participants
  Study Disease | 0
  Study Drug Toxicity: Cardiac arrest | 1
  Study Drug Toxicity: Infection with neutropenia | 1
  Study Drug Toxicity: Neutropenic sepsis | 2
  Myocardial infarction | 1

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the date of enrollment to the first date of documented disease progression or death from any cause. Because the median was not reached, results are presented as the Outcome: Number of Participants with Disease Progression or Death at Various Timepoints.
Time Frame: baseline to measured progressive disease or death from any cause (up to 68 months)
Population: Median was not reached.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the date of enrollment to the date of death from any cause. Because the median was not reached, results will be presented as the Outcome: Number of Participants who Died from Any Cause at Various Timepoints.
Time Frame: baseline to date of death from any cause up to 68 months
Population: Median was not reached
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from study enrollment to the first observation of disease progression, death as a result of any cause, or early discontinuation of treatment. Time to treatment failure was censored at the date of the last follow-up visit for patients who did not discontinue early, who were still alive, and who have not progressed. Because the upper limit of the 95% Confidence Interval of median survival was not calculable, results are presented as the Outcome: Number of Participants with Time to Treatment Failure at Various Timepoints.
Time Frame: baseline to stopping treatment (up to 68 months)
Population: Upper limit of 95% Confidence Interval of median survival was not calculable.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Patients Eligible for Breast Conservation Surgery at Baseline and Number of Patients Undergoing Breast Conservation Surgery
Description: The extent and type of surgery was guided by the tumor size, physician and/or patient decision. It was either conservation surgery or mastectomy with axillary lymph node dissection. Results are reported on the number of patients who underwent breast conservation surgery.
Time Frame: baseline, after eight 21-day cycles of study drug
Measure: Number; unit: participiants
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Number analyzed (Participants) | 65
participiants
  Eligible for Surgery at Baseline | 0
  Underwent Surgery | 18

7. Post Hoc Outcome: Number of Participants With Progressive Disease or Death at Various Time Points Throughout the Study
Description: The cumulative number of participants with an event (either progressive disease or death) are presented at various time points, as well as the number of participants at risk for the event. Participants at risk are the number of participants without progressive disease or still alive at the beginning of each time point.
Time Frame: baseline up to 68 months
Population: Intent to treat population.
Measure: Number; unit: participants
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Number analyzed (Participants) | 65
participants
  3 Months: Number of Patients with Event | 5
  3 Months: Number of Patients at Risk | 59
  6 Months: Number of Patients with Event | 8
  6 Months: Number of Patients at Risk | 50
  12 Months: Number of Patients with Event | 11
  12 Months: Number of Patients at Risk | 41
  24 Months: Number of Patients with Event | 15
  24 Months: Number of Patients at Risk | 36
  48 Months: Number of Patients with Event | 21
  48 Months: Number of Patients at Risk | 23
  68 Months: Number of Patients with Event | 21
  68 Months: Number of Patients at Risk | 1

8. Post Hoc Outcome: Number of Participants Who Died From Any Cause at Various Time Points
Description: The cumulative number of participants with an event (death from any cause) are presented at various time points, as well as the number of participants at risk for the event. Participants at risk are the number of participants still alive at the beginning of each time point.
Time Frame: baseline up to 68 months
Population: Intent to treat population.
Measure: Number; unit: participants
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Number analyzed (Participants) | 65
participants
  3 Months: Number of Patients With Event | 3
  3 Months: Number of Patients at Risk | 60
  6 Months: Number of Patients With Event | 5
  6 Months: Number of Patients at Risk | 51
  12 Months: Number of Patients With Event | 7
  12 Months: Number of Patients at Risk | 43
  26 Months: Number of Patients With Event | 11
  26 Months: Number of Patients at Risk | 37
  48 Months: Number of Patients With Event | 14
  48 Months: Number of Patients at Risk | 24
  68 Months: Number of Patients With Event | 15
  68 Months: Number of Patients at Risk | 1

9. Post Hoc Outcome: Number of Participants With Time to Treatment Failure at Various Time Points
Description: This outcome is in place of the time to treatment failure outcome. The cumulative number of participants with an event (disease progression, death as a result of any cause, or early discontinuation of treatment) are presented at various time points, as well as the number of participants at risk for the event. Participants at risk are the number of participants without disease progression, are alive, or did not discontinue treatment early at the beginning of each time point.
Time Frame: baseline to stopping treatment (up to 68 months)
Population: Intent to treat population.
Measure: Number; unit: participants
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Number analyzed (Participants) | 65
participants
  3 Months: Number of Patients with Event | 11
  3 Months: Number of Patients at Risk | 59
  6 Months: Number of Patients with Event | 19
  6 Months: Number of Patients at Risk | 50
  12 Months: Number of Patients with Event | 25
  12 Months: Number of Patients at Risk | 41
  24 Months: Number of Patients with Event | 29
  24 Months: Number of Patients at Risk | 36
  48 Months: Number of Patients with Event | 35
  48 Months: Number of Patients at Risk | 23
  68 Months: Number of Patients with Event | 35
  68 Months: Number of Patients at Risk | 1

ADVERSE EVENTS:
Arm/Group | Gemcitabine+Doxorubicin+Cisplatin+Surgery
Serious Adverse Events (participants affected / at risk) | 17/65
Other Adverse Events (participants affected / at risk) | 64/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine+Doxorubicin+Cisplatin+Surgery (N=65)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Neutropenic infection (Infections and infestations) | 2 (2)
Neutropenic sepsis (Infections and infestations) | 6 (6)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine+Doxorubicin+Cisplatin+Surgery (N=65)
Anaemia (Blood and lymphatic system disorders) | 57 (75)
Leukopenia (Blood and lymphatic system disorders) | 42 (81)
Neutropenia (Blood and lymphatic system disorders) | 45 (148)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (21)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 13 (16)
Vomiting (Gastrointestinal disorders) | 13 (17)
Asthenia (General disorders) | 11 (14)
Fatigue (General disorders) | 15 (16)
Pyrexia (General disorders) | 7 (7)
Alanine aminotransferase increased (Investigations) | 26 (33)
Aspartate aminotransferase increased (Investigations) | 27 (32)
Blood alkaline phosphatase increased (Investigations) | 9 (12)
Blood creatinine increased (Investigations) | 5 (5)
Weight decreased (Investigations) | 10 (11)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 9 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 13 (17)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days